CLINICAL TRIAL: NCT05576051
Title: Epidemiology and Efficacy of TNFi Combination Therapy (MTX+TNFi), TNFi Monotherapy, Tofacitinib Combination Therapy and Tofacitinib Monotherapy
Brief Title: To Estimate the Efficacy of Treatment With TNFi as Monotherapy or Combination Therapy With MTX and Compare and Contrast Efficacy With Tofacitinib as Monotherapy and Combination Therapy in a Real World Setting.
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A3921422
Record Dates: First submitted 2022-10-07; First posted 2022-10-12 (Actual); Results first posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- All TNFi initiations
  Interventions: Other: patterns of use of combination therapy and monotherapy
- TNFi initiations after 11/6/2012 for comparisons with Tofacitinib initiators
  Interventions: Other: patterns of use of combination therapy and monotherapy
- RA patient in Corrona with initiation Tofacitinib during follow-up in Corron
  Interventions: Other: patterns of use of combination therapy and monotherapy

INTERVENTIONS:
Other: patterns of use of combination therapy and monotherapy

SUMMARY:
To estimate the efficacy of treatment with TNFi as monotherapy or combination therapy with MTX and compare and contrast efficacy with Tofacitinib as monotherapy and combination therapy in a real world setting.

ELIGIBILITY:
Inclusion Criteria:

* RA patients in Corrona initiating a TNFi biologic (adalimumab, etanercept, infliximab, golimumab, certolizumab pegol) during follow-up in Corrona with no prior use of Tofacitinib

Exclusion Criteria:

* Patients with no history of cDMARD but history of 1+ biologics - these cases will be excluded from analyses
* Patients using combination therapy with a cDMARD other than MTX will be excluded
* Patients using combination therapy of MTX and another cDMARD will be excluded

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Observational retrospective data using the Corrona RA Registry
Sampling Method: Non-Probability Sample
Enrollment: 9159 (Actual)
Dates: Start 2015-06-04 (Actual); Primary Completion 2015-10-07 (Actual); Study Completion 2015-10-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data from greater than (>) 5500 participants who initiated Tumor Necrosis Factor Inhibitor (TNFi) initiation as combination with Methotrexate (MTX) and >2000 participants who initiated TNFi initiations as monotherapy; > 500 participants who initiated Tofacitinib initiations as monotherapy or as combination with MTX were observed in this non-interventional observational study.
Pre-assignment Details: Participants diagnosed with rheumatoid arthritis (RA), enrolled in Corrona US-based observational RA registry were included in this study.
Groups:
- All Tumor Necrosis Factor Inhibitor (TNFi) Initiators Combination: Participants diagnosed with RA, enrolled in Corrona RA registry who initiated TNFi initiators treatment with combination of MTX were included in this reporting group. Data was collected for this study from 4-Jun-2015.
- All TNFi Initiators Monotherapy: Participants diagnosed with RA, enrolled in Corrona RA registry who initiated TNFi initiators monotherapy treatment were included in this reporting group. Data was collected for this study from 4-Jun-2015.
- TNFi Initiators After 11/6/2012 Combination: Participants diagnosed with RA, enrolled in Corrona RA registry who initiated TNFi initiators treatment with combination of MTX on or after 6 November 2012 were included in this reporting group. Data was collected for this study from 4-Jun-2015.
- TNFi Initiators After 11/6/2012 Monotherapy: Participants diagnosed with RA, enrolled in Corrona RA registry who initiated TNFi initiators monotherapy treatment on or after 6 November 2012 were included in this reporting group. Data was collected for this study from 4-Jun-2015.
- Tofacitinib Initiators Combination: Participants diagnosed with RA, enrolled in Corrona RA registry who initiated Tofacitinib initiators treatment with combination of MTX were included in this reporting group. Data was collected for this study from 4-Jun-2015.
- Tofacitinib Initiators Monotherapy: Participants diagnosed with RA, enrolled in Corrona RA registry who initiated Tofacitinib initiators monotherapy treatment were included in this reporting group. Data was collected for this study from 4-Jun-2015.
Period: Overall Study
Arm/Group | All Tumor Necrosis Factor Inhibitor (TNFi) Initiators Combination | All TNFi Initiators Monotherapy | TNFi Initiators After 11/6/2012 Combination | TNFi Initiators After 11/6/2012 Monotherapy | Tofacitinib Initiators Combination | Tofacitinib Initiators Monotherapy
Started | 5077 | 2275 | 987 | 494 | 124 | 202
Completed | 4215 | 1724 | 825 | 394 | 86 | 147
Not Completed | 862 | 551 | 162 | 100 | 38 | 55
Not completed — Lack of Efficacy | 543 | 343 | 108 | 72 | 28 | 50
Not completed — Safety | 78 | 74 | 16 | 14 | 4 | 5
Not completed — Efficacy + Safety | 10 | 7 | 3 | 0 | 0 | 0
Not completed — Other | 231 | 127 | 35 | 14 | 6 | 0

BASELINE CHARACTERISTICS:
Population: Analysis population included all eligible participants whose data were observed in this study.
Groups:
- All TNFi Initiators Combination: Participants diagnosed with RA, enrolled in Corrona RA registry who initiated TNFi initiators treatment with combination of MTX were included in this reporting group. Data was collected for this study from 4-Jun-2015.
- Total: Total of all reporting groups
Arm/Group | All TNFi Initiators Combination | All TNFi Initiators Monotherapy | TNFi Initiators After 11/6/2012 Combination | TNFi Initiators After 11/6/2012 Monotherapy | Tofacitinib Initiators Combination | Tofacitinib Initiators Monotherapy | Total
Number analyzed (Participants) | 4056 | 1716 | 838 | 406 | 96 | 145 | 7257
Age, Continuous [Median (Inter-Quartile Range); unit: Years] — Population: Here, "Number Analyzed" signifies number of participants evaluable for specified arms.
  Years
    All TNFi initiators combination: number analyzed (Participants) | 4056 | 0 | 0 | 0 | 0 | 0 | 4056
    All TNFi initiators combination | 56 [48 to 65] |  |  |  |  |  | 56 [48 to 65]
    All TNFi initiators monotherapy: number analyzed (Participants) | 0 | 1716 | 0 | 0 | 0 | 0 | 1716
    All TNFi initiators monotherapy |  | 55 [46 to 63] |  |  |  |  | 55 [46 to 63]
    TNFi initiators after 11/6/2012 combination: number analyzed (Participants) | 0 | 0 | 838 | 0 | 0 | 0 | 838
    TNFi initiators after 11/6/2012 combination |  |  | 58 [50 to 66] |  |  |  | 58 [50 to 66]
    TNFi initiators after 11/6/2012 monotherapy: number analyzed (Participants) | 0 | 0 | 0 | 406 | 0 | 0 | 406
    TNFi initiators after 11/6/2012 monotherapy |  |  |  | 55 [46 to 64] |  |  | 55 [46 to 64]
    Tofacitinib initiators combination: number analyzed (Participants) | 0 | 0 | 0 | 0 | 96 | 0 | 96
    Tofacitinib initiators combination |  |  |  |  | 59 [53 to 67] |  | 59 [53 to 67]
    Tofacitinib initiators monotherapy: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 145 | 145
    Tofacitinib initiators monotherapy |  |  |  |  |  | 59 [52 to 66] | 59 [52 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3121 | 1354 | 653 | 330 | 76 | 118 | 5652
  Male | 935 | 362 | 185 | 76 | 20 | 27 | 1605
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 256 | 110 | 71 | 28 | 6 | 14 | 485
  Not Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3800 | 1606 | 767 | 378 | 90 | 131 | 6772
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 50 | 14 | 16 | 5 | 1 | 1 | 87
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 268 | 98 | 56 | 28 | 4 | 7 | 461
  White | 3389 | 1454 | 675 | 335 | 84 | 118 | 6055
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 349 | 150 | 91 | 38 | 7 | 19 | 654
History of Cardiovascular disease [Count of Participants; unit: Participants] | 306 | 139 | 69 | 32 | 8 | 16 | 570
History of cancer excluding nonmelanoma skin cancer [Count of Participants; unit: Participants] | 194 | 84 | 32 | 14 | 6 | 11 | 341
History of Diabetes [Count of Participants; unit: Participants] | 300 | 150 | 74 | 39 | 9 | 16 | 588
Smoker [Count of Participants; unit: Participants]
  Never smoker | 2084 | 864 | 388 | 195 | 49 | 78 | 3658
  Previous smoker | 1163 | 514 | 267 | 127 | 33 | 45 | 2149
  Current smoker | 787 | 327 | 172 | 77 | 13 | 21 | 1397
  Unknown or not reported | 22 | 11 | 11 | 7 | 1 | 1 | 53
Work Status [Count of Participants; unit: Participants]
  Full Time | 1697 | 672 | 331 | 150 | 29 | 41 | 2920
  Part time | 412 | 160 | 89 | 44 | 7 | 10 | 722
  Work at home | 424 | 190 | 62 | 35 | 17 | 12 | 740
  Student | 73 | 34 | 45 | 20 | 1 | 4 | 177
  Retired | 526 | 298 | 110 | 73 | 15 | 33 | 1055
  Disabled | 884 | 345 | 191 | 79 | 24 | 40 | 1563
  Unknown or not reported | 40 | 17 | 10 | 5 | 3 | 5 | 80
Insurance [Count of Participants; unit: Participants]
  None | 96 | 42 | 28 | 20 | 0 | 0 | 186
  Private | 3059 | 1293 | 609 | 296 | 62 | 112 | 5431
  Medicaid | 242 | 110 | 45 | 32 | 5 | 8 | 442
  Medicare | 1054 | 454 | 237 | 114 | 38 | 49 | 1946

OUTCOME MEASURES:

1. Primary Outcome: Clinical Disease Activity Index (CDAI) Score at 6 Months for Tofacitinib Monotherapy vs Tofacitinib With Methotrexate (MTX)
Description: CDAI was a simplified index for assessing the disease activity comprising of the swollen joint counts (SJC), tender/painful joint counts (TJC), participant's global assessment of disease activity (PtGA) and physician's global assessment of disease activity (PGA). CDAI is the numerical sum of 4 outcome parameters: SJC and TJC (based on 28-joint assessment range from 0 to 28, higher scores indicated worse condition), PtGA and PGA (score range from 0 to 10, assessed on 0-10 centimeter (cm) visual analog scale (VAS); higher scores indicated greater affection due to disease activity). CDAI total score = 0 (no disease) to 76 (severe disease), higher scores indicated worse condition. In this outcome measure, CDAI for all and non-switchers participants was reported.
Time Frame: At month 6 follow up visit
Population: Analysis population included all eligible participants whose medical records were retrieved and observed in this study. Here, "Number Analyzed (n)" signifies number of participants evaluable for specified rows.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tofacitinib Initiators Combination | Tofacitinib Initiators Monotherapy
Number analyzed (Participants) | 96 | 145
Units on a scale
  All | 18.1 (15.1) | 17 (13.4)
  Non-switchers: number analyzed (Participants) | 83 | 112
  Non-switchers | 16.6 (14.3) | 14.6 (11.6)

2. Secondary Outcome: CDAI Score at 6 Months for Tumor Necrosis Factor Inhibitor (TNFi) Monotherapy vs TNFi Combination With MTX
Description: as for outcome 1
Time Frame: At month 6 follow up visit
Population: Analysis population included all eligible participants whose medical records were retrieved and observed in this study. Here, "n" signifies number of participants evaluable for specified rows. Due to change in planned analysis, data for TNFi initiators after 11/6/2012 combination and monotherapy arms were not evaluable for CDAI score outcome measure as CDAI score data were not available in medical records for any participant in TNFi initiators after 11/6/2012 combination and monotherapy arms.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | All TNFi Initiators Combination | All TNFI Initiators Monotherapy
Number analyzed (Participants) | 4056 | 1716
Units on a scale
  All | 13.9 (12.5) | 16.5 (13.8)
  Non-switchers: number analyzed (Participants) | 3601 | 1414
  Non-switchers | 13 (11.8) | 14.9 (13)

3. Secondary Outcome: CDAI Score at 6 Months for Tofacitinib Monotherapy vs TNFi Combination With MTX
Description: as for outcome 1
Time Frame: At month 6 follow up visit
Population: Analysis population included all eligible participants whose medical records were retrieved and observed in this study. Here, "Number Analyzed" signifies number of participants evaluable for specified rows.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | All TNFi Initiators Combination | Tofacitinib Initiators Monotherapy
Number analyzed (Participants) | 4056 | 145
Units on a scale
  All | 13.9 (12.5) | 17 (13.4)
  Non-switchers: number analyzed (Participants) | 3601 | 112
  Non-switchers | 13 (11.8) | 14.6 (11.6)

4. Secondary Outcome: CDAI Score at 6 Months for Tofacitinib Combination With MTX vs TNFi Monotherapy
Description: as for outcome 1
Time Frame: At month 6 follow up visit
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | All TNFI Initiators Monotherapy | Tofacitinib Initiators Combination
Number analyzed (Participants) | 1716 | 96
Units on a scale
  All | 16.5 (13.8) | 18.1 (15.1)
  Non-switchers: number analyzed (Participants) | 1414 | 83
  Non-switchers | 14.9 (13) | 16.6 (14.3)

5. Secondary Outcome: CDAI Score at 6 Months for Tofacitinib Combination With MTX vs TNFi Combination With MTX
Description: as for outcome 1
Time Frame: At month 6 follow up visit
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | All TNFi Initiators Combination | Tofacitinib Initiators Combination
Number analyzed (Participants) | 4056 | 96
Units on a scale
  All | 13.9 (12.5) | 18.1 (15.1)
  Non-switchers: number analyzed (Participants) | 3601 | 83
  Non-switchers | 13 (11.8) | 16.6 (14.3)

6. Secondary Outcome: CDAI Score at 6 Months for Tofacitinib Monotherapy vs TNFi Monotherapy
Description: as for outcome 1
Time Frame: At month 6 follow up visit
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | All TNFI Initiators Monotherapy | Tofacitinib Initiators Monotherapy
Number analyzed (Participants) | 1716 | 145
Units on a scale
  All | 16.5 (13.8) | 17 (13.4)
  Non-switchers: number analyzed (Participants) | 1414 | 112
  Non-switchers | 14.9 (13) | 14.6 (11.6)

7. Secondary Outcome: Number of Participants With Modified American College of Rheumatology 20% (mACR20) at 6 Months for Tofacitinib Monotherapy vs Tofacitinib With MTX
Description: mACR20 response: >= 20 percent (%) improvement in tender and swollen joint count and 20% improvement in 2 of the following 4 criteria: 1) participant assessment of pain (scored from 0 to 100, higher scores indicated worsened pain) ; 2) participant global assessment of disease activity (scored from 0 to 100, higher scores indicated worsened condition); 3) physician global assessment of disease activity (scored from 0 to 100, higher scores indicated worsened condition); 4) self-assessed disability index of the mHAQ (scored from 0 to 3, higher scores indicated worsened function).
Time Frame: At month 6 follow up visit
Population: Analysis population included all eligible participants whose medical records were retrieved and observed in this study. Here, "Overall number of Participants Analyzed (N)" signifies number of participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib Initiators Combination | Tofacitinib Initiators Monotherapy
Number analyzed (Participants) | 90 | 135
Participants | 19 | 28

8. Secondary Outcome: Number of Participants With mACR20 at 6 Months for TNFi Monotherapy vs TNFi Combination With MTX
Description: as for outcome 7
Time Frame: At month 6 follow up visit
Population: Analysis population included all eligible participants whose medical records were retrieved and observed in this study. Here, "N" signifies number of participants evaluable for this outcome measure. Due to change in planned analysis, data for TNFi initiators after 11/6/2012 combination and monotherapy arms were not evaluable for mACR20 outcome measure as mACR20 data were not available in medical records for any participant in TNFi initiators after 11/6/2012 combination and monotherapy arms.
Measure: Count of Participants; unit: Participants
Arm/Group | All TNFi Initiators Combination | All TNFI Initiators Monotherapy
Number analyzed (Participants) | 4013 | 1683
Participants | 1224 | 394

9. Secondary Outcome: Number of Participants With mACR20 at 6 Months for Tofacitinib Monotherapy vs TNFi Combination With MTX
Description: as for outcome 7
Time Frame: At month 6 follow up visit
Population: Analysis population included all eligible participants whose medical records were retrieved and observed in this study. Here, "Overall number of Participants Analyzed" signifies number of participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | All TNFi Initiators Combination | Tofacitinib Initiators Monotherapy
Number analyzed (Participants) | 4013 | 135
Participants | 1224 | 28

10. Secondary Outcome: Number of Participants With mACR20 at 6 Months for Tofacitinib Monotherapy vs TNFi Monotherapy
Description: as for outcome 7
Time Frame: At month 6 follow up visit
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | All TNFI Initiators Monotherapy | Tofacitinib Initiators Monotherapy
Number analyzed (Participants) | 1683 | 135
Participants | 394 | 28

11. Secondary Outcome: Number of Participants With mACR20 at 6 Months for Tofacitinib Combination With MTX vs TNFi Combination With MTX
Description: as for outcome 7
Time Frame: At month 6 follow up visit
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | All TNFi Initiators Combination | Tofacitinib Initiators Combination
Number analyzed (Participants) | 4013 | 90
Participants | 1224 | 19

12. Secondary Outcome: Number of Participants With mACR20 at 6 Months for Tofacitinib Combination With MTX vs TNFi Monotherapy
Description: as for outcome 7
Time Frame: At month 6 follow up visit
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | All TNFI Initiators Monotherapy | Tofacitinib Initiators Combination
Number analyzed (Participants) | 1683 | 90
Participants | 394 | 19

13. Secondary Outcome: Number of Participants According to Line of Therapy at TNFi Initiation
Description: Line of therapy: 1st line: no prior use of any Disease-modifying anti-rheumatic drug (DMARD) at time of initiation. 2nd line: prior use of at least one convention DMARD (cDMARD) and no prior use of any biologic. 3rd line: prior use of at least one cDMARD and prior use of 1 biologic. 4th line: prior use of at last one cDMARD and prior use of 2 or more biologics. Number of 1st line, 2nd line, 3rd line, and 4th line of therapy was reported in this outcome measure.
Time Frame: At baseline
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | All TNFi Initiators Combination | All TNFI Initiators Monotherapy
Number analyzed (Participants) | 5077 | 2275
Participants
  1st line | 203 | 89
  2nd line | 2109 | 616
  3rd line | 1088 | 581
  4th line | 656 | 430
  Missing | 1021 | 559

14. Secondary Outcome: Number of Participants According to Line of Therapy at TNFi Initiation After 11/6/2012
Description: Line of therapy: 1st line: no prior use of any DMARD at time of initiation. 2nd line: prior use of at least one convention cDMARD and no prior use of any biologic. 3rd line: prior use of at least one cDMARD and prior use of 1 biologic. 4th line: prior use of at last one cDMARD and prior use of 2 or more biologics. Number of participants according to line of therapy at TNFi initiation after 11/6/2012 was reported in this outcome measure.
Time Frame: At baseline
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | TNFi Initiators After 11/6/2012 Combination | TNFI Initiators After 11/6/2012 Monotherapy
Number analyzed (Participants) | 987 | 745
Participants
  1st line | 54 | 361
  2nd line | 388 | 123
  3rd line | 212 | 118
  4th line | 184 | 143
  Missing | 149 | 0

15. Secondary Outcome: Number of Participants According to Line of Therapy at Tofacitinib Initiation
Description: Line of therapy: 1st line: no prior use of any DMARD at time of initiation. 2nd line: prior use of at least one convention cDMARD and no prior use of any biologic. 3rd line: prior use of at least one cDMARD and prior use of 1 biologic. 4th line: prior use of at last one cDMARD and prior use of 2 or more biologics. Number of participants according to line of therapy at tofacitinib initiation was reported in this outcome measure.
Time Frame: At baseline
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib Initiators Combination | Tofacitinib Initiators Monotherapy
Number analyzed (Participants) | 124 | 202
Participants
  1st line | 6 | 12
  2nd line | 12 | 12
  3rd line | 11 | 22
  4th line | 67 | 99
  Missing | 28 | 57

16. Secondary Outcome: Median CDAI Score at Baseline- TNFi Initiator
Description: CDAI was a simplified index for assessing the disease activity comprising of the swollen joint counts (SJC), tender/painful joint counts (TJC), participant's global assessment of disease activity (PtGA) and physician's global assessment of disease activity (PGA). CDAI is the numerical sum of 4 outcome parameters: SJC and TJC (based on 28-joint assessment range from 0 to 28, higher scores indicated worse condition), PtGA and PGA (score range from 0 to 10, assessed on 0-10 centimeter (cm) visual analog scale (VAS); higher scores indicated greater affection due to disease activity). CDAI total score = 0 (no disease) to 76 (severe disease), higher scores indicated worse condition. Baseline was defined as the time of initiation of TNFi Initiator.
Time Frame: At baseline
Population: Analysis population included all eligible participants whose medical records were retrieved and observed in this study.
Measure: Median (Inter-Quartile Range); unit: Units on a scale
Arm/Group | All TNFi Initiators Combination | All TNFI Initiators Monotherapy
Number analyzed (Participants) | 4056 | 1716
Units on a scale | 18.6 [10.1 to 29.3] | 19.7 [10.5 to 29.9]
Statistical Analysis 1: Comparison: All TNFi Initiators Combination vs All TNFI Initiators Monotherapy; Test type: Other; p = 0.278, Mixed model linear regression; Mixed model linear regression with propensity-score matched pairs as the random effect

17. Secondary Outcome: Median CDAI Score at Baseline- Tofacitinib Initiator
Description: CDAI was a simplified index for assessing the disease activity comprising of the swollen joint counts (SJC), tender/painful joint counts (TJC), participant's global assessment of disease activity (PtGA) and physician's global assessment of disease activity (PGA). CDAI is the numerical sum of 4 outcome parameters: SJC and TJC (based on 28-joint assessment range from 0 to 28, higher scores indicated worse condition), PtGA and PGA (score range from 0 to 10, assessed on 0-10 centimeter (cm) visual analog scale (VAS); higher scores indicated greater affection due to disease activity). CDAI total score = 0 (no disease) to 76 (severe disease), higher scores indicated worse condition. Baseline was defined as the time of initiation of Tofacitinib Initiator.
Time Frame: At baseline
Population: Analysis population included all eligible participants whose medical records were retrieved and observed in this study.
Measure: Median (Inter-Quartile Range); unit: Units on a scale
Arm/Group | Tofacitinib Initiators Combination | Tofacitinib Initiators Monotherapy
Number analyzed (Participants) | 96 | 145
Units on a scale | 22.1 [10.6 to 33.1] | 19 [10 to 28.3]
Statistical Analysis 1: Comparison: Tofacitinib Initiators Combination vs Tofacitinib Initiators Monotherapy; Test type: Other; p = 0.131, Mixed model linear regression; Mixed model linear regression with propensity-score matched pairs as the random effect

18. Secondary Outcome: Median CDAI Score at Baseline- TNFi Initiator After 11-6-2012
Description: CDAI was a simplified index for assessing the disease activity comprising of the swollen joint counts (SJC), tender/painful joint counts (TJC), participant's global assessment of disease activity (PtGA) and physician's global assessment of disease activity (PGA). CDAI is the numerical sum of 4 outcome parameters: SJC and TJC (based on 28-joint assessment range from 0 to 28, higher scores indicated worse condition), PtGA and PGA (score range from 0 to 10, assessed on 0-10 centimeter (cm) visual analog scale (VAS); higher scores indicated greater affection due to disease activity). CDAI total score = 0 (no disease) to 76 (severe disease), higher scores indicated worse condition. Baseline was defined as the time of initiation of TNFi initiator after 11-6-2012.
Time Frame: At baseline
Population: Analysis population included all eligible participants whose medical records were retrieved and observed in this study.
Measure: Median (Inter-Quartile Range); unit: Units on a scale
Arm/Group | TNFi Initiators After 11/6/2012 Combination | TNFI Initiators After 11/6/2012 Monotherapy
Number analyzed (Participants) | 838 | 406
Units on a scale | 19.5 [11.5 to 30.5] | 21 [12 to 30]
Statistical Analysis 1: Comparison: TNFi Initiators After 11/6/2012 Combination vs TNFI Initiators After 11/6/2012 Monotherapy; Test type: Other; p = 0.987, Mixed model linear regression; Mixed model linear regression with propensity-score matched pairs as the random effect

19. Secondary Outcome: Number of Participants According to Prior Biologic for Line of Therapy of Prior Biologics (Restricted to 3+ Line of Therapy: Prior Use of at Least One Biologic) Use at TNFi Initiation
Description: Number of participants according to prior biologic for line of therapy of prior biologics (restricted to 3+ line of therapy: prior use of at least one biologic) use at TNFi initiation was reported in this outcome measure. Line of therapy: 1st line: no prior use of any Disease-modifying anti-rheumatic drug (DMARD) at time of initiation. 2nd line: prior use of at least one convention DMARD (cDMARD) and no prior use of any biologic. 3rd line: prior use of at least one cDMARD and prior use of 1 biologic. 4th line: prior use of at last one cDMARD and prior use of 2 or more biologics.
Time Frame: At baseline
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Groups:
- All TNFi Initiators Combination(Restricted to 3+Line of Therapy: Prior Use of at Least One Biologic): Participants diagnosed with RA, enrolled in Corrona RA registry who initiated TNFi initiators treatment with combination of MTX were included in this reporting group. Data was collected for this study from 4-Jun-2015.
- All TNFI Initiators Monotherapy(Restricted to 3+Line of Therapy: Prior Use of at Least One Biologic): Participants diagnosed with RA, enrolled in Corrona RA registry who initiated TNFi initiators monotherapy treatment were included in this reporting group. Data was collected for this study from 4-Jun-2015.
Arm/Group | All TNFi Initiators Combination(Restricted to 3+Line of Therapy: Prior Use of at Least One Biologic) | All TNFI Initiators Monotherapy(Restricted to 3+Line of Therapy: Prior Use of at Least One Biologic)
Number analyzed (Participants) | 2341 | 1396
Participants
  Adalimumab | 975 | 634
  Etanercept | 1286 | 872
  Infliximab | 707 | 434
  Golimumab | 7 | 12
  Certolizumab pegol | 137 | 99
  Abatacept | 295 | 265
  Rituximab | 145 | 89
  Tocilizumab | 76 | 74
  Anakinra | 85 | 52

20. Secondary Outcome: Number of Participants According to Prior Biologic for Line of Therapy of Prior Biologics (Restricted to 3+ Line of Therapy: Prior Use of at Least One Biologic) Use at TNFi Initiation After 11/6/2012
Description: Number of participants according to prior biologic for line of therapy of prior biologics (restricted to 3+ line of therapy (LOT): prior use of at least one biologic) use at TNFi initiation after 11/6/2012 was reported in this outcome measure.
Time Frame: At baseline
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Groups:
- TNFi Initiators After 11/6/2012 Combination(Restricted to 3+LOT:Prior Use of at Least One Biologic): Participants diagnosed with RA, enrolled in Corrona RA registry who initiated TNFi initiators treatment with combination of MTX on or after 6 November 2012 were included in this reporting group. Data was collected for this study from 4-Jun-2015.
- TNFI Initiators After 11/6/2012 Monotherapy(Restricted to 3+LOT: Prior Use of at Least One Biologic): Participants diagnosed with RA, enrolled in Corrona RA registry who initiated TNFi initiators monotherapy treatment on or after 6 November 2012 were included in this reporting group. Data was collected for this study from 4-Jun-2015.
Arm/Group | TNFi Initiators After 11/6/2012 Combination(Restricted to 3+LOT:Prior Use of at Least One Biologic) | TNFI Initiators After 11/6/2012 Monotherapy(Restricted to 3+LOT: Prior Use of at Least One Biologic)
Number analyzed (Participants) | 517 | 331
Participants
  Adalimumab | 233 | 176
  Etanercept | 246 | 194
  Infliximab | 147 | 93
  Golimumab | 7 | 12
  Certolizumab pegol | 60 | 33
  Abatacept | 110 | 100
  Rituximab | 42 | 28
  Tocilizumab | 45 | 56
  Anakinra | 6 | 7

21. Secondary Outcome: Number of Participants According to Prior Biologic for Line of Therapy of Prior Biologics (Restricted to 3+ Line of Therapy: Prior Use of at Least One Biologic) at Tofacitinib Initiation
Description: Number of participants according to prior biologic for line of therapy of prior biologics (restricted to 3+ line of therapy: prior use of at least one biologic) use at tofacitinib initiation was reported in this outcome measure.
Time Frame: At baseline
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Groups:
- Tofacitinib Initiators Combination(Restricted to 3+Lineoftherapy:Prior Use of at Least One Biologic): Participants diagnosed with RA, enrolled in Corrona RA registry who initiated Tofacitinib initiators treatment with combination of MTX were included in this reporting group. Data was collected for this study from 4-Jun-2015.
- Tofacitinib Initiators Monotherapy(Restricted to 3+Lineoftherapy:Prior Use of at Least One Biologic): Participants diagnosed with RA, enrolled in Corrona RA registry who initiated Tofacitinib initiators monotherapy treatment were included in this reporting group. Data was collected for this study from 4-Jun-2015.
Arm/Group | Tofacitinib Initiators Combination(Restricted to 3+Lineoftherapy:Prior Use of at Least One Biologic) | Tofacitinib Initiators Monotherapy(Restricted to 3+Lineoftherapy:Prior Use of at Least One Biologic)
Number analyzed (Participants) | 110 | 187
Participants
  Adalimumab | 72 | 109
  Etanercept | 61 | 123
  Infliximab | 41 | 82
  Golimumab | 0 | 0
  Certolizumab pegol | 29 | 42
  Abatacept | 58 | 105
  Rituximab | 35 | 41
  Tocilizumab | 40 | 60
  Anakinra | 6 | 12

ADVERSE EVENTS:
Time Frame: Not applicable as adverse events and all-cause mortality were not planned to be evaluated for the study.
Description: Due to non-interventional nature of the study and nature of data sources, the minimum criteria for reporting an adverse event (that is, identifiable participant, identifiable reporter, a suspect product, and event) could not be met, hence adverse events were not planned to be evaluated (thus at risk appears "0").
Arm/Group | All TNFi Initiators Combination | All TNFi Initiators Monotherapy | TNFi Initiators After 11/6/2012 Combination | TNFi Initiators After 11/6/2012 Monotherapy | Tofacitinib Initiators Combination | Tofacitinib Initiators Monotherapy
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.